CLINICAL TRIAL: NCT03676374
Title: A Placebo-controlled Trial With Prucalopride for the Treatment of Typical Reflux Symptoms in Patients With Gastro-esophageal Reflux Disease With Incomplete Proton Pump Inhibitor Response
Brief Title: Prucalopride Treatment for Refractory Gastro-esophageal Reflux Disease
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Principal Investigator, Prof Dr Jan Tack, Prof. Dr., Universitaire Ziekenhuizen KU Leuven
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: S61035
Record Dates: First submitted 2018-04-10; First posted 2018-09-18 (Actual); Last update posted 2019-12-05 (Actual); Status verified 2019-12

CONDITIONS: GERD
MeSH Terms: conditions — Gastroesophageal Reflux | interventions — prucalopride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prucalopride (Experimental): Prucalopride 2mg once a day as add-on for PPI 2x/d
  Interventions: Drug: Prucalopride
- Placebo (Placebo Comparator): Placebo once a day as add-on for PPI 2x/d
  Interventions: Drug: Placebo Oral Tablet

INTERVENTIONS:
Drug: Prucalopride — Prucalopride 2mg taken once a day as add-on to PPI (2x/d)
  Arms: Prucalopride
Drug: Placebo Oral Tablet — Placebo tablet taken once a day as add-on to PPI (2x/d)
  Arms: Placebo

SUMMARY:
Up to date there is no placebo-controlled trial to investigate the effect of prucalopride in patients with proven refractory GERD. Therefore, to evaluate the efficacy of prucalopride on the improvement in symptom severity and reflux parameters, we will conduct a randomized, parallel, placebo-controlled, single-blind study. 60 patients with refractory GERD symptoms will receive either placebo or prucalopride (Resolor®) 2 mg for a period of 4 weeks. Symptom severity will be assessed by a validated reflux questionnaire (ReQuest) and reflux parameters (acid exposure time and number of reflux episodes) will be assessed by means of a 24 hour impedance-pH monitoring.

ELIGIBILITY:
Inclusion Criteria:

1. 18 to 65 years old.
2. Patients must have proven reflux, documented either by the presence of esophagitis (≥ grade B) at upper endoscopy ("on" PPI b.i.d.) in the 24 months prior to inclusion or pathological reflux parameters (acid exposure time >4% or number of reflux episodes >40) on a 24 hour impedance-pH monitoring ("on" PPI b.i.d.) in the 6 months prior to inclusion.
3. History of typical GERD symptoms during PPI treatment, at least 3 times per week for 12 weeks.
4. Daily intake of PPI treatment 12 weeks prior to inclusion, with at least 8 weeks of b.i.d. therapy (at least 2*20mg of omeprazole or equivalent).
5. Sexually active women of child bearing potential participating in the study must use a medically acceptable form of contraception. Medically acceptable forms of contraception do not include oral contraceptives, due to expected diarrhea as side effect of prucalopride. Injectable or implantable methods, intrauterine devices, or properly used barrier contraception are acceptable forms of contraception.
6. Subjects must be capable of understanding and be willing to provide signed and dated written voluntary informed consent before any protocol-specific screening procedures are performed.

Exclusion Criteria:

1. Systemic diseases, known to affect esophageal motility.
2. Colitis ulcerosa, Crohn's disease, toxic megacolon.
3. Have a cardiovascular disease or QT c>450 ms
4. Severely decreased kidney function.
5. Severely decreased liver function.
6. Surgery in the thorax or in the upper part of the abdomen (appendectomy and cholecystectomy are allowed).
7. Number of stools >3 per day.
8. Major psychiatric disorder.
9. Treatment with prucalopride prior to the start of the study.
10. Concomitant use of medications such as: anticholinergics, baclofen or prokinetics.
11. Significant neurological, respiratory, hepatic, renal, hematological, cardiovascular, metabolic or gastrointestinal cerebrovascular disease as judged by the investigator.
12. Absence of PPI intake for at least 2 consecutive days in the 2 weeks prior to the screening.
13. Pregnancy or breast feeding.
14. History of poor compliance. History of/or current psychiatric illness that would interfere with ability to comply with protocol requirements or give informed consent.
15. History of alcohol or drug abuse that would interfere with ability to comply with protocol requirements.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-02-18 (Actual); Primary Completion 2021-04 (Estimated); Study Completion 2021-04 (Estimated)

PRIMARY OUTCOMES:
change in acid exposure time | 4 weeks
  change in acid exposure time assessed by 24 hour impedance-pH monitoring.

SECONDARY OUTCOMES:
change in number of reflux episodes | 4 weeks
  change in number of reflux episodes assessed by 24 hour impedance-pH monitoring
Change in symptom severity | 4 weeks
  change in symptom severity assessed by a validated reflux questionnaire (ReQuest questionnaire and diaries)

CONTACTS AND LOCATIONS:
Locations (1):
- UZ Leuven, Leuven, Belgium